CLINICAL TRIAL: NCT05311319
Title: Hepatic Artery Infusion Chemotherapy(HAIC) Combined With Anlotinib and TQB2450 as Adjuvant Therapy in HCC Patients at High Risk of Recurrence After Resection
Brief Title: HAIC Combined With Anlotinib and TQB2450 as Adjuvant Therapy in HCC Patients With High Risk of Recurrence After Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-GZWK-03
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Hepatocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC+Anlotinib (4 Cycles) +TQB2450 (4 Cycles) (Experimental): HAIC treatment was performed one month after surgery, and Anlotinib and TQB2450 for 4 cycles.
  Interventions: Drug: HAIC+TQB2450+Anlotinib
- HAIC+Anlotinib (8 Cycles) +TQB2450 (4 Cycles) (Experimental): HAIC treatment was performed one month after surgery, and Anlotinib for 8 cycles and TQB2450 for 4 cycles.
  Interventions: Drug: HAIC+TQB2450+Anlotinib

INTERVENTIONS:
Drug: HAIC+TQB2450+Anlotinib — HAIC: FOLFOX for 24hour perfusion chemotherapy. Anlotinib: 10mg orally daily on day 1 to 14 of a 21-day cycle. TQB2450: 1200 milligrams (mg) administered intravenously (IV) on Day 1 of each 21-day cycle.

SUMMARY:
This is a single center, non-randomized, open, multi-cohort clinical, exploratory Phase II study, to evaluate the efficacy and safety of HAIC combined with TQB2450 and anlotinib as adjuvant therapy in hepatocellular carcinoma (HCC) patients at high risk of recurrence after resection.

DETAILED DESCRIPTION:
The high incidence of HCC recurrence following liver resection is a serious issue. However, no adjuvant therapy has been widely recognized at present. Interventional therapy and systemic drug therapy are common treatment methods and effective treatment for liver cancer. The combination of multiple drugs may reduce the recurrence in HCC patients with high-risk recurrence. TQB2450 is a humanized monoclonal antibody of programmed death-ligand1 (PD-L1), enabling T cells to restore immune activity and thus enhance the immune response. Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) for tumor angiogenesis and proliferative signaling.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status (ECOG-PS): 0-1;
2. The expected survival is more than 3 months;
3. Histologically or cytologically diagnosed as HCC;
4. After hepatectomy, satisfy any of the following recurrence factors: a) microvascular invasion (MVI); b) Single tumor diameter ≥ 8cm; c) The tumor grew infiltratively, unclear boundary and no complete capsule; d) Multiple tumor nodules ≥3, or nodules<3 but the diameter of a single tumor is > 3cm; e) With portal vein, hepatic vein or cholangiocarcinoma thrombus; f) tumor ruptured or invaded adjacent organs before surgery.
5. hepatitis B virus (HBV) DNA<2000IU/mL;
6. Liver function status Child-Pugh grade A (≤6);
7. The main organs function well.
8. Laboratory inspection met the following criteria: Hemoglobin (Hb) ≥8.0 g/L, Neutrophils (ANC) ≥ 1.5×10^9/L, Platelet count (PLT) ≥ 60×10^9/L, Total bilirubin (TBIL) ≤3.0 mg/dL, albumin≥28 g/L, Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase≤ 5.0 ×upper limit of normal, International Prothrombin Standardization Ratio (INR) ≤ 2.3, Thyroid-stimulating hormone (TSH) ≤upper limit of normal;
9. The woman patients of childbearing age who must agree to take contraceptive methods during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.
10. Voluntary participation and written informed consent;

Exclusion Criteria:

1. History of another malignancy tumor , except for the cured skin basal cell carcinoma and cervical carcinoma in situ)
2. Other adjuvant therapy after surgery, such as targeted drugs, programmed death-1 (PD-1) antibody and other immunotherapy, FOLFOX systemic chemotherapy;
3. The imaging examination showed residual tumor after the surgical resection;
4. Patients with previous liver transplantation or preparation for liver transplantation.
5. Patients who are allergic to components of TQB2450 and anlotinib or pharmaceutical excipients;
6. Received any live attenuated vaccine within 4 weeks of admission or during the study period;
7. Patients with a history of immunodeficiency (or autoimmune disease), or other acquired congenital immunodeficiency diseases.
8. Hypertension which cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg).
9. A history of gastrointestinal bleeding within 3 months before enrollment;
10. A history of arterial and venous thrombotic events within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
11. Hereditary or acquired hemorrhagic and thrombotic tendencies, such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.
12. Pts need to long-term anticoagulant therapy;
13. Participated in any other drug clinical studies within 3 months before enrollment;
14. A history of psychotropic substance abuse or drug abuse;
15. Patients with concomitant diseases which could seriously endanger their own safety or could affect the completion of the study according to investigators' judgment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 24 months
  DFS defined as the time from date of randomization until the date of recurrence or death due to any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  OS defined as the time from date of randomization until the date of death due to any cause
Time to recurrence (TTR) | 24 months
  TTR defined as the time from date of randomization until the date of recurrence.
Safety: adverse events | 24 months
  adverse events (AEs) categorized by severity in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China